CLINICAL TRIAL: NCT06837805
Title: Iowa Produce Prescription Program: Improving the Health Status of Iowans Facing Nutrition Insecurity
Brief Title: Iowa Produce Prescription Program
Acronym: I-PPP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Lyndi Buckingham-Schutt, Assistant Professor, Iowa State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-314
Record Dates: First submitted 2025-02-11; First posted 2025-02-20 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus Type 2; Pre-diabetes
Keywords: produce prescription; behavioral nutrition intervention; online nutrition education; self determination theory
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- I-PPP+PYP Group (Experimental): The I-PPP+PYP participants will participate in both the Iowa Produce Prescription Program and the Produce Your Path Behavioral Nutrition Intervention. This group will complete the monthly PYP intervention modules to receive the produce prescription dollar amount, which can be redeemed at partnering retail locations on fresh fruits and vegetables. An optional Facebook group for the I-PPP+PYP participants with offer additional social support and resources for participants, who can use the Facebook page to post questions, share goals and recipes, and answer prompts posted by the research team.
  Interventions: Other: Iowa Produce Prescription Program (I-PPP); Behavioral: Produce Your Path Behavioral Nutrition Intervention (PYP)
- PYP Alone Group (Experimental): The PYP Alone Group will complete the six-month behavioral nutrition intervention, but will not receive monthly incentives to redeem for fresh fruits and vegetables. PYP Alone participants will still complete the corresponding quizzes to monthly education modules. The PYP Alone participants will also have access to separate optional Facebook group to post questions, share goals and recipes, and answer prompts posted by the research team.
  Interventions: Behavioral: Produce Your Path Behavioral Nutrition Intervention (PYP)
- Control Group (No Intervention): This group will not receive the produce prescription incentive or behavioral intervention.

INTERVENTIONS:
Other: Iowa Produce Prescription Program (I-PPP) — The I-PPP intervention offers a produce prescription in the form of $30.00 per family member in a household every month to spend on fruit and vegetables. The dollars can be used at local retail partners, which are specific to each community. A mobile app has been developed for the I-PPP intervention participants. At the beginning of each month for six months, the app asks participants to complete a nutrition education module and a corresponding short quiz. After the participant completes the module, $30.00 per family member in the house will be loaded into the app for participants to use over the next month at local retail partners to buy fresh fruits and vegetables. Participants will have 30 days from the date of distribution to spend the funds before they expire.
  Arms: I-PPP+PYP Group
Behavioral: Produce Your Path Behavioral Nutrition Intervention (PYP) — The PYP Intervention is a six-month virtual behavioral intervention grounded in Self Determination Theory. The intervention aims to improve participants' competence, autonomy, and sense of relatedness through educational videos, recipes, and supplemental resources. Each monthly module contains several short videos, totaling around 15 minutes in length. The module topics include goal-setting, planning meals, preparing fruits and vegetables, reading nutrition labels, budgeting for healthier eating, and making healthier food swaps. The videos are tailored to represent a variety of cultures, ethnicities, and backgrounds, with diverse actors and recipes. Upon completion of each monthly module, a short quiz is administered to participants to measure self-efficacy related to the topic and prompt goal-setting. To further increase social support, an optional Facebook Group component allows participants to post questions, share goals and recipes, and answer prompts from the research team.
  Arms: I-PPP+PYP Group; PYP Alone Group

SUMMARY:
The goal of this study is to understand how a Produce Prescription Program paired with a behavioral nutrition intervention affect nutrition and overall health in low-income Iowans with type 2 diabetes or pre-diabetes. Research questions include:

1. What impact does a produce prescription program paired with a behavioral nutrition intervention on nutrition security compared to the behavioral nutrition intervention alone and usual care groups?
2. What impact does a produce prescription program paired with a behavioral nutrition intervention on hemoglobin A1c, fruit and vegetables intake, food security, and related behaviors compared to the behavioral nutrition intervention alone and usual care groups?

Participants of the behavioral nutrition intervention (Produce Your Path) alone will:

* Watch monthly nutrition education videos about topics like planning and budgeting for groceries, reading nutrition labels, eating more fruits and vegetables, and new recipes to try
* Complete a short quiz about their own goals and habits related to the topic
* (Optional): Join a Facebook group to communicate with other participants about their goals, share ideas and recipes, and ask questions

Participants of both the Produce Prescription and Produce Your Path Interventions will:

* Complete each monthly nutrition education module and monthly quiz
* (Optional): Join a Facebook group to communicate with other participants about their goals, share ideas and recipes, and ask questions
* Receive $30.00 per each person in their household monthly to buy fresh fruits and vegetables

Participants of the control group will:

* Follow their usual care for health conditions
* Complete the required data collection for the study

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Pre-diabetic or diabetic diagnosis by medical provider;
* Receiving medical assistance under a state plan (Medicaid) or eligible for Supplemental Nutrition Assistance Program (SNAP) benefits;
* Owns a smart phone;
* Able to read and understand English; speaks English;
* Patient at a partnering health care clinic;
* No one else in the household is enrolled in I-PPP

Exclusion Criteria:

* Under 18 years old;
* Not pre-diabetic or diabetic (as diagnosed by medical provider);
* Does not receive medical assistance under a state plan (Medicaid) or is not eligible for SNAP benefits;
* Does not own a smart phone;
* Cannot read or understand English;
* Does not speak English;
* Is not a patient at a partnering health care clinic;
* Others in household participating in I-PPP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Nutrition Security | From Month 1 of the intervention to the end of the intervention (Month 6)
  The USDA's definition of Nutrition Security is 'all Americans have consistent and equitable access to healthy, safe, affordable foods essential to optimal health and well-being'. To measure participant's nutrition security, the investigators will administer the four-item Household Nutrition Security tool developed by the Center for Nutrition & Health Impact. Participants of every arm of the study will complete the nutrition security items as part of the Baseline Survey (Month 1) and Post-Survey (Month 6). Participants will answer the four questions using a 5-point Likert frequency scale (never to always). The answers correspond to a number, and the overall score is the mean of the four answers, with lower scores indicating less nutrition security.

SECONDARY OUTCOMES:
Hemoglobin A1c (HA1c) | From Month 1 of the intervention to the end of the intervention (Month 6)
  Participant's hemoglobin A1c levels (HA1c) will be measured to help identify how well blood sugar levels are being managed. The Hemoglobin A1c test measures what percentage of blood hemoglobin proteins are glycated, with higher percentages indicating poorer glucose control and prediabetes or diabetes. This test is conducted by participant's primary care providers and data is released to the research team. HA1c will be collected from lab draws in electronic medical records.
Dietary Intake | From Month 1 of the intervention to the end of the intervention (Month 6)
  Investigators will measure participant's fruit and vegetable consumption using the 10-item dietary assessment tool from the Center for Nutrition, which was previously adapted from the Dietary Screener Questionnaire from developed by NIH and the National Cancer Insititute. The assessment tool asks participants how often they consumed certain fruits, vegetables, and food products over the last 30 days. This dietary assessment tool is part of the Baseline Survey (Month 1) and Post-Survey (Month 6).
Psychosocial Mediators | From Month 1 of the intervention to the end of the intervention (Month 6)
  Psychosocial constructs including self-efficacy, social support, and motivation level are measured in the Baseline Survey (Month 1) and Post-Survey (Month 6). Self-efficacy and social support are measured using a two- and three-item tool recommended by the Center for Nutrition, respectively. Motivational level is measured using the 15-item Treatment Self-Regulation Questionnaire, which was specifically developed to measure how intrinsically motivated a person is, as proposed by Self Determination Theory. These psychosocial constructs were chosen because the intervention is designed to increase self-efficacy and social support, and is also grounded in Self Determination Theory, aiming to increase intrinsic motivation.

OTHER OUTCOMES:
Body Mass Index (BMI) | From Month 1 of the intervention to the end of the intervention (Month 6)
  BMI from height and weight will be collected near the beginning and conclusion of the intervention by the primary care provider.
Food Security | From Month 1 of the intervention to the end of the intervention (Month 6)
  Food Security will be measured using the 6-item shortened version of the USDA's household food security tool, as recommended by the Center for Nutrition. Food security is defined as 'access by all people at all times to enough food for an active, healthy life.'
Lipid Panel | From Month 1 of the intervention to the end of the intervention (Month 6)
  Participant's serum lipids (Total cholesterol, HDL, LDL, and triglycerides) will be collected near the beginning and conclusion of the intervention by the primary care provider.
Blood Pressure | From Month 1 of the intervention to the end of the intervention (Month 6)
  The primary care provider will collect blood pressure near the beginning and conclusion of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Iowa State University, Ames, Iowa, United States

REFERENCES:
- See also: Iowa Healthiest State Initiative's Iowa Produce Rx webpage. — https://www.iowahealthieststate.com/produce-rx